CLINICAL TRIAL: NCT00771355
Title: In Vivo Imaging of Pigmentary Disorders by Reflectance Confocal Microscopy
Status: Terminated | Type: Observational
Why Stopped: Lack of study staff.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Ernesto Gonzalez, Massachusetts General Hospital
Other Study IDs: 2008-P-001137/1
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Vitiligo; Melasma; Hyperpigmentation; Hypopigmentation
MeSH Terms: conditions — Vitiligo; Melanosis; Hyperpigmentation; Hypopigmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Subjects with vitiligo.
- 2: Subjects with melasma.
- 3: Subjects with post-inflammatory hyper-pigmentation.
- 4: Subjects with post-inflammatory hypo-pigmentation.

SUMMARY:
This is a pilot study to evaluate the findings of the Reflectance Confocal Microscopy when performed in cutaneous pigmentary disorders, such as vitiligo, melasma, post-inflammatory hyper-pigmentation and hypo-pigmentation. Confocal Microscopy is a recent diagnostic technique that has been used for observation of skin conditions that affect the superficial layers of the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 20-70 years of age.
2. Clinical diagnosis of vitiligo, melasma, post-inflammatory hypo or depigmentation or post-inflammatory hyperpigmentation.
3. Willing and able to understand and sign informed consent.
4. Able to complete study and comply with study procedures.

Exclusion Criteria:

1. Use of topical therapies such as corticosteroids, protopic, hydroquinone and azelaic acid within the past 2 months.
2. Use of light therapy such as narrow-band-UVB, PUVA or laser within the past 2 months.
3. Intake of medications that can cause pigmentary changes within the past year. Examples are:

   * Antimalarials (chloroquine, hydroxychloroquine)
   * Chemotherapeutics (bleomycin, busulfan, doxorubicin, daunorubicin, fluorouracil, cyclophosphamide, and carmustine)
   * Heavy metals (gold, silver, bismuth, and mercury)
   * Tetracyclines (including minocycline, doxycycline)
   * Amiodarone
   * Azidothymidine
   * Clofazimine
4. Clinically significant abnormal findings or conditions (other than the pigmentary disorder), which might, in the opinion of the Principal Investigator, interfere with study evaluations or pose a risk to subject safety during the study.
5. Subjects who are known to be pregnant or planning a pregnancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 20-70 years of age with the clinical diagnosis of vitiligo, melasma, post-inflammatory hypo or depigmentation or post-inflammatory hyperpigmentation will be recruited from Dermatology practice at the Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
To describe characteristic features seen by confocal microscopy of several pigmentary disorders. | study visit

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Gonzalez, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rajadhyaksha M, Grossman M, Esterowitz D, Webb RH, Anderson RR. In vivo confocal scanning laser microscopy of human skin: melanin provides strong contrast. J Invest Dermatol. 1995 Jun;104(6):946-52. doi: 10.1111/1523-1747.ep12606215. PMID 7769264